CLINICAL TRIAL: NCT04963634
Title: Research of Biomarkers Associated With the Diagnosis and Severity of Bradykinin Angioedema
Acronym: BRADYDIAG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_59; 2020-A03306-33 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2021-06-02; First posted 2021-07-15 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Angio Edema
Keywords: Angioedema; Bradykinin; Biomarker; Biobanking
MeSH Terms: conditions — Angioedema | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with bradykinin angioedema
  Interventions: Other: Biobanking
- Patients with histamine-mediated angioedema
  Interventions: Other: Biobanking

INTERVENTIONS:
Other: Biobanking — For patients included in BRADYDIAG study, 2 blood samples will be collected at enrollment (for group 1: bradykinin angioedema and for group 2: histamine-mediated angioedema) and at 1 year visit (for group 1 only: bradykinin angioedema).
  Other Names: Biobanking without genetic analysis

SUMMARY:
The unpredictable nature of the attacks is one of the essential characteristics of bradykinin angioedema. The two main difficulties for physicians managing a patient with bradykinin angioedema are to make the diagnosis and anticipate the severity.

Biomarkers can be used to diagnose, guide treatment, or predict the severity of a disease. However, the identification of biomarkers is currently difficult in bradykinin both for diagnosis and prognosis. While measurement of C4 and C1 inhibitor (quantitative and functional assays) allows the diagnosis of bradykinin angioedema due to C1 inhibitor deficiency, whether genetic or acquired, many patients with normal C1 inhibitor bradykinin angioedema, either hereditary or acquired, are still difficult to diagnose. For patients with hereditary angioedema with C1-inhibitor deficiency, there is no biomarker currently available to predict the severity. Any biomarker that could improve the diagnosis on the one hand, and improve the prediction of the frequency and severity of the response to treatment on the other hand, would obviously be extremely useful. The aim of our study is to assess the existence possible biomarkers for diagnosis and prognosis of bradykinin angioedema.

ELIGIBILITY:
Inclusion Criteria:

* Group 1 : Patients with bradykinin angioedema
* Patient with biologically proven hereditary angioedema with C1 inhibitor deficiency,
* Or a patient with bradykinin angioedema related to a plasminogen or factor XII mutation,
* Or patients with bradykinin angioedema related to ACE inhibitors or ARB2,
* Or patient with acquired bradykinin angioedema due to C1 inhibitor deficiency,
* Age > or = 18 years with the capacity to understand the requirements of the study and to give a non-opposition
* Having a blood collection scheduled as part of routine care
* Being insured by social security

Group 2 : Patients with histamine-mediated angioedema

* Patient with idiopathic histamine angioedema as determined by the referring physician
* Age > or = 18 years with the capacity to understand the requirements of the study and to give a non-opposition
* Having a blood collection scheduled as part of routine care
* Being insured by social security

Exclusion Criteria:

* Minors or protected adults,
* Pregnant or breastfeeding woman,
* Person deprived of liberty,
* Person in an emergency situation,
* Person having refused or unable to give their non-opposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with bradykinin angioedema or histamine-mediated angioedema followed in internal medicine department of Lille University Hospital
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2022-01-22 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
compare measurement by proteomics of proteins differentially expressed in the plasma by ANOVA t test | through study completion an average of 1 year
  to evaluate the contribution of a plasma proteomic signature including albumin, gammaglobulin and alpha macroglobulin the plasma proteome of two group: Enrollment (for group 1 and group 2) + 1 year visit (for group 1 only)

SECONDARY OUTCOMES:
analyze the following biomarkers for diagnostic purposes in both groups. | Enrollment (for group 1 and group 2) + 1 year visit (for group 1 only)
  analyze the following biomarkers for diagnostic purposes: C1 inhibitor quantity
the value of plasma proteome markers and the markers mentioned above as predictors of the occurrence of attacks | at 1 year
Implementation of a biobank to identify future biomarkers | Enrollment (for group 1 and group 2) + 1 year visit (for group 1 only)

CONTACTS AND LOCATIONS:
Overall Officials: David Launay, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chu Lille, Lille, France